CLINICAL TRIAL: NCT01378078
Title: Transcranial Direct Current Stimulation (tDCS) for Treatment of Negative Syndrome in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Daniel Keeser, Ph.D., Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04/2011
Record Dates: First submitted 2011-06-16; First posted 2011-06-22 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Schizophrenia
Keywords: schizophrenia; negative syndrome; PANSS
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- sham (Sham Comparator): patients receive sham tDCS stimulation
  Interventions: Device: eldith DC-stimulator (neuroconn, Ilmenau, Germany)
- active (Active Comparator): active transcranial direct current stimulation
  Interventions: Device: eldith DC-stimulator (Neuroconn, Ilmenau, Germany)

INTERVENTIONS:
Device: eldith DC-stimulator (neuroconn, Ilmenau, Germany) — daily tDCS treatment over left DLPFC, 20 min, 2 mA
  Arms: sham
Device: eldith DC-stimulator (Neuroconn, Ilmenau, Germany) — same as sham stimulation
  Arms: active

SUMMARY:
Transcranial direct current stimulation (tDCS) showed beneficial effects on cognition in healthy subjects and depressed patients. In this study, patients with treatment resistant negative syndrome in schizophrenia will be treated with direct current stimulation. fMRI measures will be performed.

ELIGIBILITY:
Inclusion Criteria:

* schizophrenic patients with a negative syndrome. PANSS > 40.

Exclusion Criteria:

* other psychiatric or neurologic diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
SANS reduction | 4 weeks after baseline
  decrease by 30%

SECONDARY OUTCOMES:
neuropsychological tests | 4 weeks after baseline
  increase in SOPT by 30% increase in TMT by 30%

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Palm, MD, Principal Investigator — Ludwig Maximilian University Munich
Locations (1):
- Klinik fuer Psychiatrie, Munich, Germany